CLINICAL TRIAL: NCT05736796
Title: Effects of Complex Training On Pain and Posture In School Going Children With Heavy Bags Packs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC/PCR&AHS/22/0733
Record Dates: First submitted 2022-12-09; First posted 2023-02-21 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Posture Disorders in Children
Keywords: Abnormal posture; Back pain; Improper backs use; Physical exercise
MeSH Terms: conditions — Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General cervical Exercise (Other): Students of this group will perform general exercises of the cervical region to strengthen the Muscles.
  Interventions: Other: General cervical Exercise
- Lumber Extension Excersie (Experimental): Lumber Extension Excersie will be done to prevent the lumber straighten.
  Interventions: Other: Lumber strengthening exercises

INTERVENTIONS:
Other: Lumber strengthening exercises — Complex Training program to Achieve the normal postural. Lumber Extension Excersie will be done to prevent the lumber straighten.
  Arms: Lumber Extension Excersie
Other: General cervical Exercise — Students of this group will perform general exercises of the cervical region to strengthen the Muscles.
  Arms: General cervical Exercise

SUMMARY:
As the issues of related to heavy bag packs are increasing with every day so the complex training program along with postural training may prove to be an effective protocol in dealing with issues

ELIGIBILITY:
INCLUSION CRITERIA:

* Children with age between 12 to 15 years.
* Children with normal BMI (5th - 85th percentile).
* Students carrying bags with 15% of body weight.

EXCLUSION CRITERIA:

* Children with any physical disability ( Spinal cord injury, Cerebral palsy, Multiple sclerosis, and Epilepsy)
* Children using single-strap bags.
* One-sided shoulder elevation.
* Children using handbags or trolley bags.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating scale. | 8 weeks
  The numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Visual Analog scale | 6weeks
  The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine. Also called VAS.
  A tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Shabna Ashraf, Principal Investigator — Riphah International University
Locations (1):
- EFA school Adalat garha branch, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No